CLINICAL TRIAL: NCT04134221
Title: A Study on Internal Carotid Artery Blood Flow Velocity in Children With Moyamoya Disease Undergoing Surgery: a Prospective Observational Study
Brief Title: Internal Carotid Artery Blood Flow in Pediatric Moyamoya Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Other Study IDs: 1910-055-106
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Carotid Artery, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound assessment — Ultrasound assessment of internal carotid artery blood flow

SUMMARY:
Little is known about how general anesthesia-induced decrease in cerebral blood flow in pediatric moyamoya pateints. We investigated this question in patients undergoing moyamoya surgery, hypothesizing that cardiorespiratory changes during this procedure would reduce cerebral perfusion.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing encephaloduroarteriosynangiosis surgery for moyamoya disease

Exclusion Criteria:

* cutaneous lesion on the neck

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric Moyamoya disease patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Internal carotid artery blood flow velocity | from anesthetic induction to end of surgery, an average of 5 hours
  ultrasound assessment of internal carotid artery blood flow velocity

CONTACTS AND LOCATIONS:
Locations (1):
- Hee-Soo Kim, Seoul, Soul-t'ukpyolsi, South Korea

IPD SHARING:
Plan to Share IPD: Undecided